CLINICAL TRIAL: NCT03439319
Title: Restoration of Reaching and Grasping Function in Individuals With Spinal Cord Injury Using MyndMove® Neuromodulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MyndTec Inc. (Industry)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Programs for Assessment of Technology in Health Research Institute (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MM-SCI-4002; CDMRP-SC150251 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs(CDMRP),Spinal Cord Injury Research Program, US Dept of Defense)
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Spinal Cord Injuries; Trauma, Nervous System
Keywords: MyndMove; Electrical neuromodulation; conventional therapy
MeSH Terms: conditions — Spinal Cord Injuries; Trauma, Nervous System

STUDY DESIGN:
Intervention Model Description: A two-arm, parallel group, multicentre, single-blind, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MyndMove® therapy (Active Comparator): Non-invasive Functional Electrical Stimulation (FES) technique with surface electrodes to stimulate from 3 to 8 muscles to create purposeful movements in one or both hands/arms
  Interventions: Device: MyndMove®
- Intensive Conventional therapy (Active Comparator): Using Conventional therapy which focuses exclusively on the purposeful movements in one or both hands/arms
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Device: MyndMove® — This FES therapy can be used as a short-term therapeutic intervention to help improve voluntary grasping function
  Arms: MyndMove® therapy
Other: Conventional Therapy — Conventional training involves repetitive practice of upper extremity movements with manual assistance provided by a therapist as needed.
  Arms: Intensive Conventional therapy

SUMMARY:
A two-arm, parallel group, multicentre, single-blind, randomized controlled trial comparing electrical neuromodulation delivered by MyndMove® therapy to intensive upper-limb conventional therapy in the treatment of patients with moderate to severe motor impairment to their arms and hands from an incomplete, traumatic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic incomplete (AIS B-D) C4-C7 spinal cord injury
2. Paralysis or paresis in both upper extremities
3. At least 4 months (120 days) and less than 96 months (2,920 days) post traumatic SCI
4. Baseline SCIM-SC ≤ 10
5. From an inpatient or outpatient care setting
6. Able to understand and follow instructions
7. Able to tolerate being in a seated position for a least one hour required to deliver upper limb therapy
8. Willing to attend treatment sessions and all assessment sessions
9. Able to understand and provide informed consent
10. Male and female participants ≥ 18 years of age at the time of enrollment

Exclusion Criteria:

1. Previous history of any other neuromuscular disorder or conditions that may affect motor response
2. Upper extremity injury or condition prior to SCI that limits the function of the hand or arm
3. Malignant skin lesion on the affected upper extremity
4. Rash or open wound at any potential electrode site
5. History of seizure disorder not effectively managed by seizure medications
6. An implanted metallic part (e.g. plates, screws or joint replacement) or electrical device (e.g. Implantable Cardiac Defibrillator, Pacemaker, Spinal Stimulation). (Note: If the participant has passive metallic implants, the therapy can be delivered if the implants are located in an area other than where the electrical stimulant is to be delivered.)
7. Complete denervation of muscles that are targeted by MyndMove such that MyndMove is unable to elicit tetanic muscle contraction when upper limits of stimulation intensity for the targeted muscle are applied
8. Poorly controlled autonomic dysreflexia (as determined by the local site physician)
9. History of psychiatric illness requiring hospitalization within the past 24 months
10. Active drug treatment for dementia
11. Life expectancy of less than 12 months due to other illness
12. In the judgment of the medical provider, the participant has medical complications that may interfere with the execution of the study
13. Currently enrolled in another upper limb study and/ or has received MyndMove Therapy within the past 3 months
14. Enrolled, in the past six months, in a clinical study involving drugs or biologics
15. Currently dependent on a ventilator
16. Botulinum toxin injection into affected upper extremity and the muscle targeted by MyndMove® therapy within 6 months prior to the study start. No botulinum toxin injections in the upper extremity during the study treatment and follow up period
17. Females who are pregnant or planning to become pregnant in the duration of the trial
18. Regional disorder of the upper extremities such as fracture, dislocation, or joint contractures to less than 50% of the expected range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of MyndMove® therapy vs intensive conventional therapy in improving upper extremity function as measured by Spinal Cord Independence Measure self-care sub score (SCIM-SC) | Change from baseline to 6weeks to 14 weeks to 24weeks
  SCIM-SC is a disability scale that has been specifically developed to evaluate the functional outcomes of patients with traumatic and non-traumatic SCI. The SCIM-SC assesses function of self-care, which includes feeding, bathing, dressing and grooming.

SECONDARY OUTCOMES:
Change in participant's upper limb and hand impairment and function using Graded Refined Assessment of Strength Sensibility and Prehension (GRASSP) | Change from baseline to 6weeks to 14weeks to 24weeks
  This is a multi-modality test designed to assess the integration of sensorimotor hand and upper limb impairment and function. This test combines the features of several other tests that have been used to assess hand and upper limb function in the peripheral hand population
Change in participant's reaching and grasping function with the Toronto Rehab Institute Hand Function Test (TRI-HFT) | Change from baseline to 14 weeks to 24weeks
  A test developed to evaluate improvements in the gross motor function of the unilateral grasp due to FES for reaching and grasping treatment. Hand functions that will be tested with the TRI-HFT are: lateral or pulp pinch, and palmar grasps.
  that have been used to assess hand and upper limb function in the peripheral hand population
To assess safety as measured by serious and non serious adverse events (SAEs) recorded for participants in both groups of the study population over the duration of the study | Duration of the trial from baseline to 24weeks
Change in quality of life as measured by the Spinal Cord Injury-Quality of Life (SCI-QOL) | Change from baseline to 6weeks to 14weeks to 24weeks
  The SCI-QOL measurement system is a multifaceted system of measuring patient reported outcomes across a wide variety of functioning specifically targeted for individuals with SCI

CONTACTS AND LOCATIONS:
Overall Officials: Steve Plymale, Study Director — MyndTec Inc.
Locations (4):
- United States (2):
  - MetroHealth Medical Center / Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - TIRR Memorial Hermann, Houston, Texas
- Canada (2):
  - HealthTech Connex Centre for Neurology Studies / NeuroMotion Physiotherapy Clinics ( Surrey, Vancouver and Victoria), Surrey, British Columbia
  - Toronto Rehabilitation Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson KD, Korupolu R, Musselman KE, Pierce J, Wilson JR, Yozbatiran N, Desai N, Popovic MR, Thabane L. Multi-center, single-blind randomized controlled trial comparing functional electrical stimulation therapy to conventional therapy in incomplete tetraplegia. Front Rehabil Sci. 2022 Sep 9;3:995244. doi: 10.3389/fresc.2022.995244. eCollection 2022. PMID 36188946
- [Derived] Anderson KD, Wilson JR, Korupolu R, Pierce J, Bowen JM, O'Reilly D, Kapadia N, Popovic MR, Thabane L, Musselman KE. Multicentre, single-blind randomised controlled trial comparing MyndMove neuromodulation therapy with conventional therapy in traumatic spinal cord injury: a protocol study. BMJ Open. 2020 Sep 28;10(9):e039650. doi: 10.1136/bmjopen-2020-039650. PMID 32988951